CLINICAL TRIAL: NCT06637449
Title: Identification of Bacterial and Fungal Isolates in Patients with Sinonasal Polyps
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Ahmed Allam Ahmed, Identification of bacterial and fungal isolates in patients with sinonasal polyps, Assiut University
Other Study IDs: Bacterial in sinonasal polyps
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Sinonasal Polyps
Keywords: Bacterial culture from patients with sinonasal polyi

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Intra-operative nasal Swab from the sinuses ( ethmoidal or maxillary ) to detect bacterial and fungal growth by using VITEK 2 ( fully automated system for microbial identification and antimicrobial susceptibility testing ) in clinical pathology department in AUH
  Equipment Details :
  Instrument: Vitek 2 Compact 30 Serial Number: VK2C14152 Software Version: V9.02
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To detect bacterial and fungal growth in patients with sinonasal polyps undergoing FESS

DETAILED DESCRIPTION:
Chronic rhinosinusitis with nasal polyps (CRSwNP) is a disease of the nose and paranasal sinuses characterized by mucosal thickening and polyp formation¹ which are inflammatory lesions that project into the nasal airway and are typically bilateral² .Chronic rhinosinsitis with nasal ployps (CRSwNP) affects 0.5% to 4% of the population worldwide. ³ Symptoms include anterior or posterior rhinorrhea, nasal congestion, hyposmia, and/or facial pressure or pain that last for a duration of more than 12 weeks.² The cause of the sinonasal polyps is still unknown but they may be associated with several pathological conditions i.e. infection, allergic fungal sinusitis, allergy and cystic fibrosis ⁴. Many studies were based on detection of bacterial and fungal growth in sinonasal polyps , and found that preoperative bacterial culture showed growth of Staphylococcus coagulase negative (CONS) ,Staphylococcus aureus , gram -ve bacteria i.e. Pseudomonas aeruginosa , Klebsiella pneumoniae , Klebsiella ozenae and Escherichia coli⁴ . From fungi , Aspergillus species were the most commonly recovered isolates ⁵. The initial approach of management was medical treatment . Medical therapy consists of administration of intranasal or systemic steroids. Other medical treatments considered the use of antibiotics, leukotriene modifiers, and avoidance of acetylsalicylic acid. Surgical removal was performed for non-responders to medical management⁶. Functional endoscopic sinus surgery (FESS) is a minimally invasive technique in which sinus air cells and sinus ostia are opened under direct visualization. The goal of this procedure is to restore ventilation and normal functions⁷.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adult patients (18 and over )

2. Patients with sinonasal polyposis confirmed with nasal endoscopy and Computed tomography and undergoing FESS

Exclusion Criteria:

* 1.Chronic rhinosinsits without nasal polyps 2. Patients below 18 years old and above 70 years old 3. Immunocompromised patient. 4. Recent administration of antibiotics or antifungal medication . 5. Unilateral nasal polyp , granuloma and tumors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with nasal polyps ,their age between 18 years to 70 years , undergoing FESS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of bacterial and fungal colanization in patients of chronic rhinosinsitis with nasal polyps | 15 days

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jain S, Das S, Gupta N, Malik JN. Frequency of fungal isolation and antifungal susceptibility pattern of the fungal isolates from nasal polyps of chronic rhinosinusitis patients at a tertiary care centre in north India. Med Mycol. 2013 Feb;51(2):164-9. doi: 10.3109/13693786.2012.694486. Epub 2012 Jul 12. PMID 22783803
- [Background] Andrews AE, Bryson JM, Rowe-Jones JM. Site of origin of nasal polyps: relevance to pathogenesis and management. Rhinology. 2005 Sep;43(3):180-4. PMID 16218510
- [Background] Stevens WW, Schleimer RP, Kern RC. Chronic Rhinosinusitis with Nasal Polyps. J Allergy Clin Immunol Pract. 2016 Jul-Aug;4(4):565-72. doi: 10.1016/j.jaip.2016.04.012. PMID 27393770
- [Background] Van Zele T, Gevaert P, Holtappels G, Beule A, Wormald PJ, Mayr S, Hens G, Hellings P, Ebbens FA, Fokkens W, Van Cauwenberge P, Bachert C. Oral steroids and doxycycline: two different approaches to treat nasal polyps. J Allergy Clin Immunol. 2010 May;125(5):1069-1076.e4. doi: 10.1016/j.jaci.2010.02.020. PMID 20451040